CLINICAL TRIAL: NCT03759509
Title: Effects of Aerobic Exercise Training on Nurses' Sleep Quality, Fatigue, Attention and Cortisol Profile: A Randomized Controlled Trial
Brief Title: Effects of Aerobic Exercise Training on Nurses' Sleep Quality, Fatigue, Attention and Cortisol Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMU-JIRBN201711007
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2018-11

CONDITIONS: Nurse; Attention; Aerobic Exercise; Sleep Quality; Fatigue; Cortisol
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will randomly sample from previously screen low sleep quality participants, then random assign to experimental (aerobic exercise) and control (routine activity) groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise training (Experimental): three times a week, a total of twenty-four times in eight weeks
  Interventions: Behavioral: aerobic exercise
- control (No Intervention): routine activity

INTERVENTIONS:
Behavioral: aerobic exercise — the experimental group, in which aerobic exercise training is given three times a week, a total of twenty-four times in eight weeks
  Arms: aerobic exercise training

SUMMARY:
Shift work in nursing has been found to result in sleep disruption and sleep deprivation, and in sleepiness or fatigue at work. Slow reaction, insufficient attention and poor judgement often come with increased fatigue, which contributes to a high risk of accident and patient safety. Studies have shown that aerobic exercise is helpful in promoting high sleep quality. The study is conducted a prospective parallel randomized trial is performed to 60 nurses with low sleep quality. The subjects are randomly assigned to: (i) the experimental group, in which aerobic exercise training is given; (ii) the control group, in which the subjects kept their original lifestyles. The study aims to investigate the effects of aerobic exercise training on nurses' sleep quality, fatigue, attention and cortisol profile.

DETAILED DESCRIPTION:
When work shifts and lifestyles change, the synchronous relationship between the body's biological clock and the environment, i.e., circadian rhythms, is disrupted, resulting in insufficient sleep and insomnia. Shift work in nursing has been found to result in sleep disruption and sleep deprivation, and in sleepiness or fatigue at work. Slow reaction, insufficient attention and poor judgement often come with increased fatigue, which contributes to a high risk of accident and patient safety. Studies have shown that aerobic exercise is helpful in promoting high sleep quality, whereas few researchers have argued over how aerobic exercise training improves sleep quality in nurses. The study is conducted in two stages. Previous stage, we conducted with a cross-sectional study design with convenience sampled 200 participants to fill out the Chinese Pittsburgh Sleep Quality Index (CPSQI) questionnaire for screen the low sleep quality (CPSQI > 5) participants. A total of 200 nurses were recruited, and 199 valid samples were collected, 108 participants were found to have low sleep quality (CPSQI > 5). The study will adopt a prospective, longitudinal, parallel-group comparative study, randomly sample from previously screen low sleep quality participants, then random assign to experimental (aerobic exercise) and control (routine activity) groups, and actigraphy sleep recording, saliva samples and attention data will be collected.

The study aims to investigate the effects of aerobic exercise training on nurses' sleep quality, fatigue, attention and cortisol profile. The findings of the study could provide guidelines on improving nurses' fitness and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Full-time
* Female nursing staff members
* Worked 8 hours per shift
* Had at least 1 year of work experience.

Exclusion Criteria:

* Had used sedatives, hypnotics, antihistamines, or hormonal drugs within the 4 weeks before commencing the study
* Pregnant
* Were diagnosed as having sleep or stress disorders, or experienced sleep problems owing to concurrent insomnia or sleep apnea.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Total sleep time sleep change | The 1st workday 8:00AM to 5th workday 8:00AM of 4th, 8th, and 12th week
  The actigraphy reported on sleep parameters of the amount of actual sleep minutes
Wake after sleep onset change | The 1st workday 8:00AM to 5th workday 8:00AM of 4th, 8th, and 12th week
  The actigraphy reported on the amount of minutes they were awake between sleep onset and wake time.
Sleep efficiency change | The 1st workday 8:00AM to 5th workday 8:00AM of 4th, 8th, and 12th week
  The actigraphy reported on sleep parameters of percentage of time asleep while in bed from lights off to lights on.
Seep onset latency change | The 1st workday 8:00AM to 5th workday 8:00AM of 4th, 8th, and 12th week
  The actigraphy reported on sleep parameters of the minutes between lights off and first sleep episode.

SECONDARY OUTCOMES:
Simple visual reaction time testing | Before and after work, the test are completed within 5 min
  Psychomotor Vigilance Task Monitor to test simple visual reaction time
Saliva cortisol | Collected at awakening [0 min] and at 30 min, 6 hours, and 12 hours after awakening
  Diurnal cortisol concentration

CONTACTS AND LOCATIONS:
Overall Officials: shu fen Niu, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No